CLINICAL TRIAL: NCT02970773
Title: Prospective, Non-randomized, Open-label, Mono-centric, Cohort Study on the Absorption of Oral Rivaroxaban in Patients With a Cervical Spinal Cord Injury
Brief Title: Absorption of Rivaroxaban in Patients With Cervical Spinal Cord Injury
Acronym: rivaroxaban
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment; sponsor-investigator has left the institution
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-21
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Spinal Cord Injuries; Thromboembolism
MeSH Terms: conditions — Spinal Cord Injuries; Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rivaroxaban (Other): Rivaroxaban Oral Tablet
  Interventions: Drug: Rivaroxaban Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban Oral Tablet — oral application of Xarelto

SUMMARY:
The primary objective of this study is to investigate the pharmacokinetic and -dynamic properties of rivaroxaban after oral administration in cervical spinal cord injury (SCI) individuals.

The secondary objective of this study is to determine the steady-state rivaroxaban activity in cervical SCI individuals under long-term therapy.

Primary Objective In-house patients will be informed concerning the study and informed consent will be collected.

During the screening day, in- / exclusion criteria will be assessed and a blood samples will be taken for assessing haematology, clinical chemistry and coagulation parameters. Furthermore, the evaluation day will be scheduled.

On the evaluation day, in- / exclusion criteria will be re-assessed. A venous catheter will be introduced into a forearm or lower leg of each participant for the collection of blood at the specified time points. Skin inspection for subcutaneous bleeding will be performed and vital signs will be recorded. A blood sample will be taken for assessing haematology, clinical chemistry and coagulation parameters.

Single administration of oral rivaroxaban in the form of Xarelto® 10mg tablets (Bayer Schering Pharma, Berlin, Germany).

Rivaroxaban concentrations will be determined from plasma samples taken before, 30min after and 1, 2, 3, 4, 5, 6, 8, 12, 24 hours after rivaroxaban administration. Rivaroxaban activity will be determined from plasma samples taken before, 30min after and 1, 2, 3, 4, 5, 6, 8, 12, 24 hours after rivaroxaban administration using a factor Xa inhibition test and measuring prothrombin time (PT) and activated partial thromboplastin time (aPTT).

Skin inspection for subcutaneous bleeding and measurements of vital signs will be performed 30min and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours after rivaroxaban administration.

Secondary Objective Patients under long-term rivaroxaban therapy will be recruited during their annual check-up visit at the Swiss Paraplegic Centre. In- / exclusion criteria will be assessed, and the patients will be informed concerning the study and informed consent will be collected.

Blood samples will be taken for assessing haematology, clinical chemistry and coagulation parameters, and skin inspection for subcutaneous bleeding and measurements of vital signs will be performed.

A blood sample (4.3ml citrated venous blood) will be taken for assessing the primary and secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Motor complete tetraplegia for at least 3 months
* Age from 18 to 74 years
* Body mass index (BMI) from 18 to 35kg/m2
* Informed consent as documented by signature

Exclusion Criteria:

* Any anti-coagulation therapy (apart from rivaroxaban for second objective)
* Hypersensitivity or allergy to factor Xa inhibitors
* Acute bacterial endocarditis
* Bleeding disorder
* Clinically relevant active bleeding
* Gastrointestinal ulcer or tumor
* Hepatic dysfunction with increased bleeding risk
* Renal failure / patients undergoing dialysis
* Pregnancy and breast feeding
* Gastrectomy, biliopancreatic diversion, resection or re-routing of small intestines
* Feeding tube
* Recent blood donation
* Abnormalities of laboratory values: alanine-aminotransferase (ALAT), aspartate-aminotransferase (ASAT), gamma-glutamyl transferase (gammaGT), alkalic phosphatase (AP), bilirubin, amylase, lipase, cystatin C, creatinine, white blood cell count, haemoglobin, platelet count, prothrombin time, aPTT, fibrinogen, thrombin time, factors II,V,VII and X
* Use of therapeutic or recreational drugs influencing plasmatic coagulation

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
rivaroxaban plasma level | before drug administration and 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h and 24h after drug administration

SECONDARY OUTCOMES:
inhibition of factor XII | before drug administration and 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h and 24h after drug administration
prothrombin time | before drug administration and 30min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h and 24h after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Felleiter, MD PhD, Principal Investigator — Swiss Parapelgic Centre
Locations (1):
- Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No